CLINICAL TRIAL: NCT03212820
Title: Clinical Evaluation of the Effect of Low Speed Drilling Versus Conventional Drilling Technique on Crestal Bone Level in Maxilla. A Randomized Controlled Clinical Trial
Brief Title: Low Speed Drilling Versus Conventional Drilling Technique on Crestal Bone Level in Maxilla.(Group B ) A Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Tarek, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cebc.cairoun
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biologic drilling (Experimental): drilling at low speed
  Interventions: Procedure: Drilling at low speed
- conventional drilling (Active Comparator): drilling at conventional or high speed
  Interventions: Procedure: Drilling at conventional or high speed

INTERVENTIONS:
Procedure: Drilling at low speed
  Arms: Biologic drilling
Procedure: Drilling at conventional or high speed
  Arms: conventional drilling

SUMMARY:
20 patients were selected requiring implant placement and divided randomly into two groups (10 in each group)

* for the study group, starter drill is used to locate the point of insertion as planned then pilot drill is also used to the full desired working length after that all other sequential drills are used at a low speed (50-70 rpm) without irrigation .
* In the study group: implant will be inserted in the low speed osteotomy site.
* In the control group: implants will be inserted in the conventional prepared osteotomy site.
* For both groups there is no surgical guide used.
* The flap will then be copiously irrigated with saline in preparation for closure.
* The flap will then be closed using interrupted 4/0 resorbable sutures.

ELIGIBILITY:
Inclusion Criteria:

* Patients restoring missing maxillary teeth with implant placement.
* Both sexes.
* Age: 25-45
* Mesio-distal dimensions: Not less than 6 mm
* Bone Height: Not less than 12 mm
* Bucco-lingual dimensions: Not less than 8mm
* All measures will be assessed using CBCT.

Exclusion Criteria:

* Sites needing bone grafting or augmentation.
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
crestal bone loss | 6 month
  measurement from radiographic analysis using digital periapical x-ray

SECONDARY OUTCOMES:
patient morbidity after procedure | 1 day
  pain value on pain scale
Implant stability value | 3 month
  resonance frequency analysis using osstell

IPD SHARING:
Plan to Share IPD: Yes